CLINICAL TRIAL: NCT02879370
Title: "Transanal Inspection and Management of Low ColoRectal Anastomosis Performed With a New Technique: the TICRANT Study"
Brief Title: Transanal Inspection and Management of Low ColoRectal Anastomosis Performed With a New Technique
Acronym: TICRANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: San Giuseppe Moscati Hospital (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Casa di Cura San Pio X, Milano, Italy (Unknown); Policlinico Abano Terme (Other); Ospedale Maggiore, Bologna Italy (Unknown)
Responsible Party: Principal Investigator, Pierpaolo Sileri, MD, PhD, FACS Assistant Professor of Surgery, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 65/14
Record Dates: First submitted 2014-11-24; First posted 2016-08-25 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Anastomotic Leak
Keywords: Anastomotic Leak; Rectal cancer; Double stapling technique
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TICRANT (Experimental): Transanal Inspection and management of low ColoRectal Anastomosis
  Interventions: Procedure: Transanal Inspection and management of low ColoRectal Anastomosis

INTERVENTIONS:
Procedure: Transanal Inspection and management of low ColoRectal Anastomosis — Low anterior resection with total mesorectal excision (TME), either performed open, laparoscopic or robotic Closure of the rectum with linear or curved stapler with transanal inspection Transanal placement of four 2-0 prolene sutures on the rectal stump, respectively 2 at the extremities of the suture line (left and right) and other two 1 cm medial to each of the previous two sutures Circular stapler is introduced, the 4 tails of the prolene stitches are introduced through the windows (2 in the left and 2 in the right side of the instrument) and gently pulled, to obtain a gradual and homogeneous traction of the tissue and elimination of both previous suture lines and doggy ears, then the stapler is fired The termino-terminal anastomosis is carefully inspected A leak test can be performed (if negative the protective stoma is not performed) An eventual leak can be transanally repaired

SUMMARY:
The technique the investigators propose to perform colorectal and colo-anal anastomosis in patients underwent low and ultra-low anterior resection for rectal cancer could potentially reduce the anastomotic leakage rate by better trans-anal introduction of the circular stapler, elimination of the previous suture lines and dog ears, combined with direct inspection of the anastomosis, easy performance of trans-anal air leak tests and eventually direct repair of any small anastomotic defects. Another important point in cancer surgery is the easily identification of the distal margin. In fact, this technique is simple to perform, reproducible and safe in terms of complications.

DETAILED DESCRIPTION:
-Study design Subjects for this study were prospectively enrolled between January 2013 and January 2016 in the participating centers.

All patients signed written informed consent including the possibility of future publication according to the Italian bioethics laws. Institutional Review Board (IRB) approval has been obtained from the local Ethical Committee of each center in compliance with the Principals of Helsinki Declaration.

-Preoperative assessment and preparation All cases were discussed individually on colorectal multidisciplinary meeting with standard preoperative staging for rectal cancer including; colonoscopy with biopsy, CT chest, and abdomen, MRI pelvis and/or endo-rectal ultrasound. All patients were evaluated preoperative by expert anesthesiologists for individual co-morbidity with classification according to the ASA score.

The day before surgery mechanical bowel preparation with 4 liters of PEG (PolyEthilene Glycol) was administered together with liquid diet. An adequate thromboembolic prophylaxis with low molecular weight heparin was given the evening before the surgery. Antibiotic prophylaxis with second generation cephalosporin was administered at induction of anesthesia.

-Surgical technique The low or ultra-low anterior resection with total mesorectal excision (TME) were performed, either open, laparoscopic, robotic. Just before rectal division, the circular anal dilator (CAD) device was introduced into the anal canal and fixed by four 0-silk suture to the perianal skin apply at the 4 cardinal's points. The rectal inspection was carried out by the Purse Suture Anoscope (PSA) to correctly identify the proximal and distal extension of the tumor. After that the rectum was divided by linear or curved stapler under CAD direct inspection.

Four 2-0 prolene sutures were trans-anally placed on the rectal stump; 2 of them at the extremities of the suture line (left and right) and the other two 1 cm medially to each of the previous two sutures. Circular stapler was introduced through the CAD (29 or 33 mm KOL stapler, Touchstone International Medical Science Co., Ltd.), the 4 tails of the prolene stitches were introduced through the stapler channels (2 in the left and 2 in the right side of the instrument) and gently pulled in order to obtain a gradual and homogeneous traction of the tissue. After elimination of both previous suture lines and dog ears, then the stapler was fired.

The rectal anastomosis was carefully inspected trans-anally then tested intraoperatively by air leak test through trans-anal air insufflation with the pelvis immersed with physiological saline to detect bubbles, and competence of donuts. If the anastomosis was considered safe the need for protective stoma was left to discretion of operating surgeon.

CAD may be removed at the end of the surgery, or left in place for 3-4 days postoperative to provide a safe and fast access for anastomosis inspection as well to reduce the endo-luminal pressure.

* Postoperative care The postoperative care concise with the standard care for patients who underwent low or ultra-low rectal resection, thromboembolic prophylaxis continued inform of single low molecular weight heparin 5000 IU 8 hours postoperative or according to the risk status of patients. Antibiotics for 3 days postoperative inform of 1 gm 2nd generation cephalosporin. We encourage fast tract surgery inform early feeding and mobilization as described below;

  * 1st POD: removal of the urinary catheter, start mobilization,
  * 2nd POD: start oral fluid,
  * 3rd-4th POD: start semi-solid then solid feeling,
  * 5-6th POD: discharge home (after performing contrast enema or colonoscopy).
* Definition of anastomotic leak There is no constant definition for anastomotic leak, but we adapted the criteria recently published by Adams and Papagrigoriadis [8]; feculent material from the drain or the wound, extravasation of dye on contrast enema, anastomotic defect visualized by colonoscopy, or the presence of peri-anastomotic air or fluid visualized by CT scan.
* Patient's fellow-up Patients were followed-up at the outpatient's clinics at one week, two weeks, and at one month postoperative. A further follow-up occurred at time of stoma reversal in patients with diversion in form of colonoscopy to access anastomotic integrity and preoperative anesthetic fitness as usual. Follow-up was continued at twelve months' postoperative by aid of complete colonoscopy.
* Variables studied and statistical analysis Basic demographic data were recorded including age and sex of patients as well as detailed information on BMI, ASA, stage and distance of the tumor from anal verge, neo-adjuvant chemotherapy, type of surgical approach (open, laparoscopic and robotic procedure), duration of the operation, postoperative hospital stay, postoperative morbidity and mortality. Data were analyzed using excel and SPSS (Statistical Package for Social Science) version 21 programs under Microsoft Windows. Quantitative data were expressed as mean ± SD when possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing low or ultra-low anterior resection for biopsy proven primary rectal cancer

Exclusion Criteria:

* Patients younger than 18 years old,
* pregnant,
* recurrent disease,
* cancer less than 4 cm from the anal verge,
* abdomeno-perineal resection,
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Incidence of anastomotic leakage after intervention | 1 year
  The authors adapted these criteria for diagnosis of anastomotic leakage; fecal material from the drain or the wound, extravasation of dye on contrast enema, anastomotic defect visualized by colonoscopy, or the presence of peri-anastomotic air or fluid visualized by CT scan.

SECONDARY OUTCOMES:
Safety margin after tumor resection | 1 year
  postoperative pathology of tumor specimen wiyh asscesment of cancer free both radial and distal margins
Postoperative morbidities and mortalities | 1 year
  Overall all deaths or complications occurred during the surgery or 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Crafa, MD, Study Director — San Giuseppe Moscati Hospital; Giovanni Romano, MD, Study Chair — Fondazione G. Pascale; Jacques Megevand, MD, Study Chair — Pavia University
Locations (1):
- University of Rome Tor Vergata, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dehni N, Schlegel RD, Cunningham C, Guiguet M, Tiret E, Parc R. Influence of a defunctioning stoma on leakage rates after low colorectal anastomosis and colonic J pouch-anal anastomosis. Br J Surg. 1998 Aug;85(8):1114-7. doi: 10.1046/j.1365-2168.1998.00790.x. PMID 9718009
- [Background] Edwards DP, Leppington-Clarke A, Sexton R, Heald RJ, Moran BJ. Stoma-related complications are more frequent after transverse colostomy than loop ileostomy: a prospective randomized clinical trial. Br J Surg. 2001 Mar;88(3):360-3. doi: 10.1046/j.1365-2168.2001.01727.x. PMID 11260099
- [Background] Heuschen UA, Hinz U, Allemeyer EH, Autschbach F, Stern J, Lucas M, Herfarth C, Heuschen G. Risk factors for ileoanal J pouch-related septic complications in ulcerative colitis and familial adenomatous polyposis. Ann Surg. 2002 Feb;235(2):207-16. doi: 10.1097/00000658-200202000-00008. PMID 11807360
- [Background] Kockerling F, Rose J, Schneider C, Scheidbach H, Scheuerlein H, Reymond MA, Reck T, Konradt J, Bruch HP, Zornig C, Barlehner E, Kuthe A, Szinicz G, Richter HA, Hohenberger W. Laparoscopic colorectal anastomosis: risk of postoperative leakage. Results of a multicenter study. Laparoscopic Colorectal Surgery Study Group (LCSSG). Surg Endosc. 1999 Jul;13(7):639-44. doi: 10.1007/s004649901064. PMID 10384066
- [Background] Marusch F, Koch A, Schmidt U, Geibetaler S, Dralle H, Saeger HD, Wolff S, Nestler G, Pross M, Gastinger I, Lippert H. Value of a protective stoma in low anterior resections for rectal cancer. Dis Colon Rectum. 2002 Sep;45(9):1164-71. doi: 10.1007/s10350-004-6384-9. PMID 12352230
- [Background] Merad F, Hay JM, Fingerhut A, Yahchouchi E, Laborde Y, Pelissier E, Msika S, Flamant Y. Is prophylactic pelvic drainage useful after elective rectal or anal anastomosis? A multicenter controlled randomized trial. French Association for Surgical Research. Surgery. 1999 May;125(5):529-35. PMID 10330942
- [Background] Moran BJ. Stapling instruments for intestinal anastomosis in colorectal surgery. Br J Surg. 1996 Jul;83(7):902-9. doi: 10.1002/bjs.1800830707. PMID 8813772
- [Background] Pakkastie TE, Ovaska JT, Pekkala ES, Luukkonen PE, Jarvinen HJ. A randomised study of colostomies in low colorectal anastomoses. Eur J Surg. 1997 Dec;163(12):929-33. PMID 9449446
- [Background] Selvasekar CR, Cima RR, Larson DW, Dozois EJ, Harrington JR, Harmsen WS, Loftus EV Jr, Sandborn WJ, Wolff BG, Pemberton JH. Effect of infliximab on short-term complications in patients undergoing operation for chronic ulcerative colitis. J Am Coll Surg. 2007 May;204(5):956-62; discussion 962-3. doi: 10.1016/j.jamcollsurg.2006.12.044. PMID 17481518
- [Background] Urbach DR, Kennedy ED, Cohen MM. Colon and rectal anastomoses do not require routine drainage: a systematic review and meta-analysis. Ann Surg. 1999 Feb;229(2):174-80. doi: 10.1097/00000658-199902000-00003. PMID 10024097
- [Background] Vignali A, Fazio VW, Lavery IC, Milsom JW, Church JM, Hull TL, Strong SA, Oakley JR. Factors associated with the occurrence of leaks in stapled rectal anastomoses: a review of 1,014 patients. J Am Coll Surg. 1997 Aug;185(2):105-13. doi: 10.1016/s1072-7515(97)00018-5. PMID 9249076
- [Background] Wexner SD, Cohen SM, Ulrich A, Reissman P. Laparoscopic colorectal surgery--are we being honest with our patients? Dis Colon Rectum. 1995 Jul;38(7):723-7. doi: 10.1007/BF02048029. PMID 7607032
- See also: The published paper — http://journals.sagepub.com/doi/10.1177/1553350617709182